CLINICAL TRIAL: NCT02298387
Title: A Phase 1 Dose Escalation and Expansion Study of OMP-305B83 in Subjects With Solid Tumors
Brief Title: A Phase 1 Study of OMP-305B83 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B83-001
Record Dates: First submitted 2014-11-10; First posted 2014-11-24 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Advanced Solid Tumor Malignancies
MeSH Terms: interventions — navicixizumab; Antibodies, Bispecific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMP-305B83 (Experimental): The dose levels of OMP-305B83 will be 0.5, 1.0, 2.5, 5 and 10 mg/kg administered IV once every 3 weeks.
  Interventions: Drug: OMP-305B83

INTERVENTIONS:
Drug: OMP-305B83 — intravenous (in the vein) infusions
  Other Names: bispecific monoclonal antibody

SUMMARY:
This is an open-label Phase 1 dose escalation and expansion study of OMP-305B83 in subjects with previously treated solid tumors. Study includes a dose escalation phase and expansion phase. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy.

DETAILED DESCRIPTION:
This is an open-label Phase 1 dose escalation and expansion study of OMP-305B83 in subjects with previously treated solid tumors. Study includes a dose escalation phase and expansion phase. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed malignancy that is metastatic or unresectable for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit or they must be ineligible to receive such therapy and/or have declined all such therapy. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT or MRI.
2. FFPE tumor tissue either fresh core needle biopsied or archived (two FFPE cores preferred whenever possible) is required for participation in the study. If fresh tissue is obtained, the core biopsy must be done at least ≥7 days prior to Day 0.
3. Subjects must have received their last chemotherapy, non-anti-VEGF biologic, or investigational therapy at least 4 weeks prior to enrollment, 6 weeks if the last regimen included BCNU or mitomycin C, and 8 weeks if the last regimen was an anti-VEGF therapy
4. Age >21 years
5. ECOG performance status <2
6. Life expectancy of more than 3 months
7. Subjects must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count >1000/mL (without a colony stimulating factor within the last 2 weeks)
   * Hemoglobin >10.5 g/dL (without erythropoietin or blood transfusion within the last 2 weeks)
   * Platelets >100,000/mL (without platelet transfusion within the last 2 weeks)
   * Total bilirubin <1.5 X institutional upper limit of normal (ULN)
   * AST (SGOT) and ALT (SGPT) <2 X institutional ULN (for subjects with hepatic metastases <5 X institutional ULN)
   * INR and PTT within 1.5 X institutional ULN
   * Proteinuria < trace
   * Creatinine <1.5 X institutional ULN OR
   * Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
8. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Subjects receiving any other investigational agents
2. Subjects who have received an anti-DLL4 antibody, or an anti-DLL4/VEGF bispecific antibody Subjects who have received prior anti-VEGF therapy are eligible, unless they have residual serious adverse events related to their anti-VEGF therapy.
3. Subjects with a history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess; clinical signs or symptoms of GI obstruction and/or requirement for parenteral hydration or nutrition. In addition, subjects with other known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease.
4. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
5. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
6. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
7. Pregnant women or nursing women
8. Subjects with known HIV infection
9. Known bleeding disorder or coagulopathy
10. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
11. Subjects with ascites or pleural effusion requiring drainage within the last 28 days.
12. Subjects with a blood pressure of >140/90 mmHg.
13. Subjects with squamous cell carcinoma of the lung
14. Subjects having undergone a major surgery within the last 6 weeks
15. New York Heart Association Classification II, III, or IV (see APPENDIX D)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Subjects will be assessed for DLTs from Days 0-21. Adverse events will be reported through 30 days after discontinuation of treatment
  Number of subjects with a DLT
Incidence of adverse events | Up to 2 years
  Number of subjects with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) - AUC, Clearance, volume of distribution, apparent half-life | PK analyses at various time points following the 1st and 3rd doses, pre-dose at Day 84 and every 9 weeks while on study, at treatment term, every 6 weeks for 12 weeks post termination
  Area under the plasma concentration-time curve, measurement of renal clearance from the body, volume of distribution, apparent half life of antibody

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD,FACP, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Oncology Research Associates, PLLC d/b/a Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma